CLINICAL TRIAL: NCT05700396
Title: Increasing Receipt of Guideline Concordant Survivorship Care Among Black Breast Cancer Survivors Through Patient Education
Brief Title: Breast Cancer Survivor Educational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Erica T. Warner, ScD MPH, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-509
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Carcinoma; Breast Cancer Female
Keywords: Breast Cancer; Breast Neoplasms; Breast Carcinoma; Breast Cancer Female; Breast cancer survivor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breast Cancer Survivor Education Program (Experimental): Participants will complete study procedures as outlined:
  - 6 weekly sessions of a modified version of the PAVING the Path to Wellness education program.
  Interventions: Behavioral: Breast Cancer Survivor Education Program

INTERVENTIONS:
Behavioral: Breast Cancer Survivor Education Program — Weekly sessions via Zoom platform with study staff.

SUMMARY:
The goal of this study is to test a 6-week virtual education program among Black breast cancer survivors. The virtual program includes sessions on physical activity, goal setting, nutrition, sleep, stress, and social connections.

DETAILED DESCRIPTION:
This six-week feasibility study will evaluate a virtual support and education program among up to 15 Black female breast cancer survivors. Participants will be asked to attend a 90 minute group session once a week for 6 weeks and complete surveys pre and post intervention surveys to ascertain study endpoints. This study is supported by funding from Pfizer and in-kind support from the American Cancer Society, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Self-identified Black or African American race
* Age 22-79
* Diagnosis of Stage I, II, or III invasive breast cancer
* Completed active treatment at least 6 months ago, but within the past five years
* Speaks English

Exclusion Criteria:

* Undergoing active treatment (i.e., surgery, chemotherapy, radiation)
* Undergoing evaluation for suspected recurrence

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment Retention Rate | 6 weeks
  Defined as the number of recruited participants who initiate intervention program.
Time Required to Recruit to Target | 6 weeks
  Defined as the amount of time to target accrual goal.
Proportion of Eligible Participants | 6 weeks
  Defined as the number of eligible participants required to recruit required sample size.
Rate of Intervention Completion | 6 weeks
  Defined as the number of participants who attend at least 5 of 6 sessions.
Success Rate of Educational Intervention | 6 weeks
  Proportion of participants "very satisfied" or "completely satisfied" with intervention. Defined successful if true of 80% of participants.
Data collection feasibility | 6 weeks
  Proportion of participants completing evaluation surveys each at baseline and week 6.

SECONDARY OUTCOMES:
Self-Efficacy for symptom self-management | 6 weeks
  Self-Efficacy for symptom self-management will be assessed using Symptom-Management Self-Efficacy Scale-Breast Cancer
Intention to Receive post-treatment Surveillance Mammography | 6 weeks
  Intention to Receive post-treatment Surveillance Mammography will be assessed using Follow-Up Care Use and Health Outcomes of Cancer Survivors (FOCUS) Survey
Physical Activity Goal Change | 6 weeks
  Physical Activity Goal Change will be assessed using Follow-Up Care Use and Health Outcomes of Cancer Survivors (FOCUS) Survey
Dietary Behavior Goal Change | 6 weeks
  Dietary Behavior Goal Change will be assessed using Follow-Up Care Use and Health Outcomes of Cancer Survivors (FOCUS) Survey
Unmet information Needs | 6 weeks
  Unmet information Needs will be assessed using Follow-Up Care Use and Health Outcomes of Cancer Survivors (FOCUS) Survey

CONTACTS AND LOCATIONS:
Overall Officials: Erica Warner, MPH, ScD, Principal Investigator — Massachusetts General Hospital; Amy Comander, MD, Study Director — Massachusetts General Hospital; Naomi Ko, MD, Study Director — Boston Medical Center
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation